CLINICAL TRIAL: NCT05210387
Title: Open-label, Randomized Clinical Trial to Assess the Non-inferiority of 7-day Antibiotic Therapy Compared to Conventional 14-day Treatment in Multidrug-resistant Gram-negative Bacilli Infections
Brief Title: Seven Versus 14 Days of Antibiotic Therapy for Multidrug-resistant Gram-negative Bacilli Infections
Acronym: OPTIMISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 47366621.1.1001.5330
Record Dates: First submitted 2021-12-31; First posted 2022-01-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-09

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection; Bloodstream Infection; Severe Infection; Pseudomonas Aeruginosa; Acinetobacter Infections; Gram-Negative Bacterial Infections; Human; Carbapenem Resistant Bacterial Infection; Bacteremia; Sepsis
MeSH Terms: conditions — Sepsis; Infections; Pseudomonas Infections; Acinetobacter Infections; Gram-Negative Bacterial Infections; Bacteremia | interventions — Duration of Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 7-day adequate antibiotic therapy (Experimental): Adequate antibiotic therapy is defined as antimicrobial treatment with at least one agent with in vitro susceptibility.
  Interventions: Other: Duration of therapy
- 14-day adequate antibiotic therapy (Active Comparator): Adequate antibiotic therapy is defined as antimicrobial treatment with at least one agent with in vitro susceptibility.
  Interventions: Other: Duration of therapy

INTERVENTIONS:
Other: Duration of therapy — In experimental group patients with severe infection caused by MDR-GNB and who present a clinical response on day 7 (±1) of adequate antimicrobial therapy, the therapy will be suspended.
  The active control group will continue therapy until day 14 (±1).

SUMMARY:
Antimicrobial resistance is a major global problem, particularly in hospital-acquired infections (HAIs). Gram-negative bacilli (GNB), including Enterobacterales, Pseudomonas aeruginosa, and Acinetobacter baumannii, are among the most common pathogens associated with multidrug resistance and HAIs. These bacteria are of special concern because few therapeutic options are available.

Traditionally, the duration of treatment for severe multidrug-resistant (MDR)-GNB infections is 14 days. Studies of severe infections by GNB, regardless of susceptibility profile, have shown that shorter antimicrobial treatments are not inferior to traditional durations of therapy and are associated with a lower incidence of adverse effects. However, there are currently no studies assessing whether shorter duration of antimicrobial treatment is effective for MDR-GNB.

This open-label, randomized clinical trial aims to assess the non-inferiority of 7-day antibiotic therapy compared to conventional 14-day treatment in severe infections by MDR-GNB.

ELIGIBILITY:
Inclusion criteria

* Infection's diagnosis while in the ICU
* Severe infection in any site (defined as the presence of sepsis/septic shock or bloodstream infection or pneumonia) associated with a positive culture by MRD-GNB (Acinetobacter baumannii complex, Pseudomonas aeruginosa, and Enterobacterales bacteria, only susceptible to carbapenems and/or polymyxins)
* Hemodynamically stable and afebrile (axillary temperature less than 37.8ºC) for at least 48 hours on day 7 of adequate antibiotic therapy
* Consent of the team providing care to the patient regarding their inclusion in the research

Exclusion criteria

* Inclusion in other experimental studies involving antimicrobial therapy
* Infections that have as the primary site: endocarditis/endovascular infection, necrotizing fasciitis, osteomyelitis, abdominal abscess or other abdominal infections requiring surgical intervention (except infections that have been treated surgically, with curative character within the first 3 days of appropriate antimicrobial therapy), central nervous system Infections, empyema, prosthetic infection;
* Immunosuppression defined as: neutrophil cells <1000/mm³ in the current hospitalization, HIV/AIDS diagnosis with last CD4 count <200/mm³, solid organ transplantation in the last year and/or need for increased immunosuppression due to acute rejection in the last year, hematopoietic stem cell transplantation in the last year, and/or current therapy for chronic graft-versus-host disease
* Positive blood cultures for the same pathogen within 48 hours prior to randomization, when collected
* Uncontrolled concomitant infection with another GNB (regardless of susceptibility profile)
* Previous inclusion in this study
* Known pregnancy
* Patient in palliative care who has already decided not to restart antimicrobials, if necessary, or hemodynamic support measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical failure | 28 days after randomization
  Incidence of clinical failure. Clinical failure is a composite outcome defined by the presence of one of the following: Infection relapse (infection anywhere in the body by the same MDR-GNB) or Death

SECONDARY OUTCOMES:
Days alive and free from hospitalization | 28 days after randomization
  Number of days in which patients are alive and out of the hospital
Days alive and free from any antibiotic therapy | 28 days after randomization
  Number of days in which patients are alive and free from any antibiotic therapy
Occurrence of infections caused by other MRD-GNB or other bacteria | 28 days after randomization
  Incidence of infections caused by other MRD-GNB or other bacteria
Length of intensive care unit stay | 28 days after randomization
  Number of days in which patients stayed at intensive care unit
Acute kidney injury | 28 days after randomization
  Incidence of acute kidney injury, according to Kidney Disease: Improving Global Outcomes (KDIGO) criteria
Diarrhea for any cause | 28 days after randomization
  Incidence of any diarrhea. Diarrhea is defined as 3 or more episodes per day.
Confirmed infection by Clostridioides difficile | 28 days after randomization
  Incidence of Clostridioides difficile infection
Hemodynamic instability lasting more than 6 hours | 14 days after randomization
  Incidence of hemodynamic instability lasting more than 6 hours. Hemodynamic instability is defined as hypotension that requires the use of doses of dopamine above 15 mcg/kg/min, epinephrine above 0.1 mcg/kg/min, or norepinephrine above 0.1 mcg/kg/min
Other adverse events related to antimicrobial therapy | 28 days after randomization
  Incidence of any other adverse event related to antimicrobial therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Prehn Zavascki, Principal Investigator — Hospital Moinhos de Vento
Locations (29):
- Brazil (29):
  - Hospital OTO clinica, Fortaleza, Ceará
  - Hospital Evangélico de Vila Velha, Vila Velha, Espírito Santo
  - Hospital Cleriston de Andrade, Feira de Santana, Estado de Bahia
  - Hospital Couto Maia, Salvador, Estado de Bahia
  - Hospital da Cidade, Salvador, Estado de Bahia
  - Instituto Hospital de Base do Distrito Federal, Brasília, Federal District
  - Hospital Universitário de Brasília, Brasília, Federal District
  - Hospital Presidente Vargas, São Luís, Maranhão
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Vila da Serra (Instituto Materno Infantil de Minas Gerais S/A), Nova Lima, Minas Gerais
  - Irmandade da Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Hospital Universitário da Universidade Estadual de Londrina, Londrina, Paraná
  - Hospital Municipal de Maringá, Maringá, Paraná
  - Hospital Regional Baixo Amazonas, Santarém, Pará
  - Hospital do Tricentenário, Olinda, Pernambuco
  - Hospital São João Batista, Volta Redonda, Rio de Janeiro
  - Hospital Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Hospital Geral Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUC, Porto Alegre, Rio Grande do Sul
  - Hospital Santa Cruz, Santa Cruz do Sul, Rio Grande do Sul
  - Hospital Ana Nery, Santa Cruz do Sul, Rio Grande do Sul
  - Hospital São Lucas Sergipe - Rede D´or São Luiz, Aracaju, Sergipe
  - Hospital Dr. Léo Orsi Bernadres - HLOB, Itapetininga, São Paulo
  - Hospital Naval Marcílio Dias, Rio de Janeiro
  - Instituto Estadual do Cérebro Paulo Niemeyer (Pró Saúde- Associação Beneficente de Assistência Social e Hospitalar), Rio de Janeiro
  - Hospital A.C Camargo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arns B, Kalil AC, Sorio GGL, Boschi E, Antonio ACP, Antonio JP, Birriel DC, Lanziotti DH, da Cunha Abbott F, Rocha GC, de Fatima Fernandes V, de Souza Dantas VC, da Silva Medeiros GF, de Franca Diniz Rocha V, Pereira FC, Gobatto ALN, Lima VP, Lacerda FH, de Maio Carrilho CMD, de Oliveira Cardozo KDN, Irineu VM, Kurtz P, Horvath JDC, Sesin GP, Agani CAJO, Dos Santos TM, Brochier LSB, da Rosa BS, Tomazini BM, Besen BAMP, Pereira AJ, Veiga VC, Nascimento GM, Zavascki AP; OPTIMISE Study Group. Seven versus 14 days of antimicrobial therapy for severe multidrug-resistant Gram-negative bacterial infections in intensive care unit patients (OPTIMISE): a randomised, open-label, non-inferiority clinical trial. Crit Care. 2024 Dec 18;28(1):412. doi: 10.1186/s13054-024-05178-6. PMID 39695798
- [Derived] Arns B, Horvath JDC, Rech GS, Sesin GP, Agani CAJO, da Rosa BS, Dos Santos TM, Brochier LSB, Cavalcanti AB, Tomazini BM, Pereira AJ, Veiga VC, Nascimento GM, Kalil AC, Zavascki AP. A Randomized, Open-Label, Non-inferiority Clinical Trial Assessing 7 Versus 14 Days of Antimicrobial Therapy for Severe Multidrug-Resistant Gram-Negative Bacterial Infections: The OPTIMISE Trial Protocol. Infect Dis Ther. 2024 Jan;13(1):237-250. doi: 10.1007/s40121-023-00897-9. Epub 2023 Dec 16. PMID 38102448